CLINICAL TRIAL: NCT00850408
Title: Enhancing the Response to Rehabilitative Interventions After Stroke Using Transcranial Magnetic Stimulation
Brief Title: Enhancing the Response to Rehabilitation After Stroke Using Repetitive Transcranial Magnetic Stimulation (rTMS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lisa Koski, PhD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 172502; CHIR MOP 84354; CHIR MOP 84354 (Other: CHIR)
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Stroke
Keywords: Stroke; rTMS; TMS; Rehabilitation; Upper Extremity
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real rTMS (Experimental): Real rTMS - subjects receiving real repetitive TMS - 1Hz over unaffected hemisphere
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham rTMS
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Procedure: Repetitive Transcranial Magnetic Stimulation — For real rTMS,1200 pulses will be delivered at a frequency of 1Hz, with an intensity equal to the 115% of the motor threshold as established at baseline. For Sham rTMS, procedures will be identical to those used for real rTMS with the exception that a placebo coil will be used, which provides acoustic and sensory stimulation like the real coil but does not stimulate neural tissue. 20-minute Real and Sham stimulation sessions will be administered bi-weekly for a period of 4 weeks

SUMMARY:
Weakness of the arm and hand results in long-term disability for many persons who suffer a stroke. After the initial recovery phase, only limited gains are achieved by retraining the weak limb to perform daily tasks. However, new treatment strategies such as repetitive transcranial magnetic stimulation (rTMS) show promise for enhancing motor recovery after stroke. rTMS is a noninvasive technique for modifying brain activity that aims to improve motor function by correcting abnormal patterns that occur after stroke. We believe that giving rTMS right before a therapy session will prepare the brain so that the patient is better able to participate in and benefit from training of the hand and arm. The goal of this study is to test how well this new strategy works to improve recovery in people who have mild to moderate weakness of the arm and hand after stroke.

Participants will receive magnetic stimulation of the movement area of the brain just prior to arm and hand training for a series of eight sessions. We will evaluate changes in hand and arm function after the intervention and one month later to see if the changes are maintained. We will also test whether some groups of people benefit more than others from the intervention. If improvements in hand and arm function are observed after the intervention, we will test it more rigourously in a future clinical trial in which participants are randomly assigned to different treatment conditions. This research will show whether brain stimulation can be used to improve the effectiveness of rehabilitation care.

ELIGIBILITY:
Inclusion Criteria:

* first clinical stroke involving the middle cerebral artery confirmed by CT or MRI scan during acute care at the MUHC, or second stroke involving the same hemisphere when there were no clinical residual effects from the first stroke;
* cortical or subcortical stroke resulting in hemiparesis;
* at least 3 months post-stroke;
* discharged from standard rehabilitation;
* able to provide informed consent, to follow instructions and participate in therapy, as evidenced by Mini Mental State Exam score > 14;
* able to understand instructions in English or French.

Exclusion Criteria:

* minimal or no residual upper extremity motor impairment;
* severe upper extremity motor impairment as indicated by inability to produce any voluntary contraction of intrinsic hand muscles; severe cognitive impairment in language or attention sufficient to impair communication during the consenting or intervention procedures (score < 14 on the Mini Mental Status Exam);
* other central nervous system disorder or peripheral neuropathy of the upper extremity;
* pain, spasticity, or other complications that would prevent participation in the intervention;
* history of seizure confirmed by interview and medical chart review;
* comorbidity such as Parkinson's disease, osteoarthritis, or cancer, precluding full participation in the assessments and in the experimental intervention;
* other conditions that increase the risk of side effects due to rTMS procedures: metal in cranium, intracardiac line, increased intracranial pressure, pregnancy, cardiac pacemaker, medication pump, tricyclic antidepressants, neuroleptics, history of seizure in the immediate family

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The Box and Blocks Test of Manual Dexterity | Post-intervention and 1 month later

SECONDARY OUTCOMES:
Cortical excitability of the motor system | Post-intervention and one month later

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Koski, PhD, Principal Investigator — McGill University
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Higgins J, Koski L, Xie H. Combining rTMS and Task-Oriented Training in the Rehabilitation of the Arm after Stroke: A Pilot Randomized Controlled Trial. Stroke Res Treat. 2013;2013:539146. doi: 10.1155/2013/539146. Epub 2013 Dec 3. PMID 24363954